CLINICAL TRIAL: NCT01079702
Title: A Phase I/II, Non-randomized, Multi-center, Dose-escalating, Two-stage Efficacy and Feasibility Study of the Combination of Everolimus and Capecitabine in Patients With Advanced Malignancies
Brief Title: Everolimus and Capecitabine in Patients With Advanced Malignancy
Acronym: m-TOR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: J.W.Wilmink, MD PhD, Academisch Medisch Centrum-Universiteit Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCmedonc08/010
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2008-01

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — Everolimus; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Everolimus — Everolimus, administrated twice daily at a fixed total dose of 10 mg continuously.
  Other Names: Certican
Drug: Capecitabine — Capecitabine administered bid for 14 days followed by 7 days rest. In this study, capecitabine will be dose escalated. The first dose level of capecitabine is 500 mg/m2 twice daily.
  Other Names: Xeloda

SUMMARY:
In the investigators study the investigators combine everolimus, administrated twice daily at a fixed total dose of 10 mg continuously with capecitabine administered bid for 14 days followed by 7 days rest. In this study, capecitabine will be dose escalated.

DETAILED DESCRIPTION:
The results form preclinical studies suggest that mTOR inhibitors are promising drugs for the treatment of various types of cancer. Everolimus seems the most attractive mTOR inhibitor because of the favourable pharmacokinetic profile and possibility of oral administration. Based on preclinical findings, mTOR inhibitors may be more efficacious when used in a rational combination with other cancer regiments like cytostatic drugs. Indeed, several multiagent combinations are being investigated in clinical trials at the moment, and the results are promising.

In our study we combine everolimus, administrated twice daily at a fixed total dose of 10 mg continuously with capecitabine administered bid for 14 days followed by 7 days rest. In this study, capecitabine will be dose escalated. The first dose level of capecitabine is 500 mg/m2 twice daily. Three patients will be enrolled per dose level, starting at dose level 1. If one of the 3 patients develops dose-limiting toxicity at any dose level, 3 other patients will start at the same dose level. If 2 or more out of these 6 patients develop DLT, no further dose escalations will be performed. The MTD will be considered to be the dose given at the previous lower level. No intrapatient dose escalation will be applied.

Once the MTD of capecitabine is established, the phase II part of the study will start in which 25 patients with various malignancies will be enrolled to evaluate the efficacy and feasibility of the combination of everolimus and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological confirmed malignancies
* Measurable lesion according to RECIST criteria (only for the phase II part of the study)
* ECOG / WHO performance status of 0-2
* Age ≥ 18 years
* Life expectancy of at least 3 months
* Minimal acceptable safety laboratory values defined as:
* WBC ≥ 3.0 x 109 /L
* Platelet count ≥ 100 x 109 /L
* Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALT or AST ≤ 2.5 x ULN, in case of liver metastases ≤ 5 x ULN
* Renal function as defined by creatinine < 150μmol/L
* Able and willing to give written informed consent
* Able to swallow and retain oral medication
* Able and willing to undergo blood sampling for pharmacokinetic and pharmacogenetic analysis
* Mentally, physically and geographically able to undergo treatment and follow up.

Exclusion Criteria:

* Patients with known alcoholism, drug addiction and/or psychotic disorders in the history that are not suitable for adequate follow up
* Women who are pregnant or breast feeding
* Women of childbearing potential who refuse to use a reliable contraceptive method throughout the study
* Serious concomitant systemic disorder that would compromise the safety of the patient, at the discretion of the investigator
* Any other medical condition that would interfere with study procedures and/or decrease safety of the protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Phase I part: Assessment of dose limiting toxicity and maximum tolerated dose. II part: efficacy and feasibility. Primary endpoint of the study will be response rate. | During treatment: assessments on day 1 every cycle (3 weeks). After treatment: every 3 months during the first 2 years, and every 6 months thereafter
  Three patients will be enrolled per dose level, starting at dose level 1. If one of the 3 patients develops dose-limiting toxicity at any dose level, 3 other patients will start at the same dose level. If 2 or more out of these 6 patients develop DLT, no further dose escalations will be performed. The MTD will be considered to be the dose given at the previous lower level. No intrapatient dose escalation will be applied.

SECONDARY OUTCOMES:
Time to treatment failure | Every 3 months during the first 2 years, and every 6 months thereafter.
Toxicity profile. | During treatment: assessments on day 1 every cycle (3 weeks). After treatment: every 3 months during the first 2 years, and every 6 months thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Wilmink, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands